CLINICAL TRIAL: NCT00771342
Title: A Blinded Placebo Controlled Single Cross-over Clinical Trial to Evaluate Fungicidal Activity With Topical Application of 1% Gaseous Nitric Oxide in Subjects With Moderate to Severe Tinea Pedis (Athlete's Foot)
Brief Title: Efficacy Study to Evaluate the Effect of Nitric Oxide on the Treatment of Tinea Pedis (Athlete's Foot)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nitric BioTherapeutics, Inc (Industry)
Responsible Party: Chief Technology Officer, Nitric BioTherapeutics, Inc.
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CTP 6
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2010-02

CONDITIONS: Tinea
MeSH Terms: conditions — Tinea | interventions — Nitric Oxide; Nitrogen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 1% gasoue nitric oxide, delivered topically for 40 minutes daily for three consecutive days
  Interventions: Drug: Nitric Oxide
- 2 (Placebo Comparator): Nitrogen gas delivered topically for 40 minutes, daily, for 3 consecutive days
  Interventions: Drug: Nitrogen

INTERVENTIONS:
Drug: Nitric Oxide — 1% gaseous nitric oxide, delivered for 40 minutes daily for 3 consecutive days
  Arms: 1
Drug: Nitrogen — Nitrogen gas, delivered topically for 40 minutes daily for 3 consecutive days
  Arms: 2

SUMMARY:
The purpose of this study is to determine the fungicidal efficacy of nitric oxide and it's effect on the clinical signs and symptoms associated with Tinea Pedis

ELIGIBILITY:
Inclusion Criteria:

* Positive clinical findings for moccasin, interdigital or bullous tinea pedis as determined by direct clinical examination
* Must have a clinical symptom severity score of at least 20 on a possible 64 point scale
* Written informed consent must be obtained from the subject.
* Must ≥ 19 years of age
* Must agree to avoid professional pedicures or application of any nail polish product or nail cosmetic to the toenails after the screening visit until the conclusion of the trial.
* Must agree to take measures to avoid pregnancy during the 12 day (or 26 day if in cross over group) study period

Exclusion Criteria:

* Has a diagnosis of either psoriasis or eczema
* Has a visual diagnosis, by the investigator, of onychomycosis.
* Use of topical antifungals e.g. (clotrimazole, ketoconazole,miconazole, oxiconazole- (Oxistat®, Glaxo Smith Kline), sulconazole, naftifine (Naftin®, Merz), terconazole, econazole nitrate (Spectazole®, Ortho-McNeil), butoconazole ,Fluconazole, ciclopirox olamine-(Loprox®, Medicis), tolnaftate, haloprogin), Zeasorb-AF , antibacterials and corticosteroids in the preceding 5 days of screening visit (Day 1)
* Use of systemic corticosteroids in the preceding 7 days of screening visit (Day 1)
* Use of systemic antifungals in the preceding 7 days of screening visit (Day1) including - (terbinafine - (Lamisil®, Novartis), Itraconazole - (Sporanox®, Janssen), fluconazole- (Diflucan®, Pfizer), ketoconazole, miconazole, griseofulvin (Gris-PEG®, Pedinol), butoconazole, terconazole, Potassium iodide)
* Has used any investigational drug(s) within 30 days preceding screening visit (Day 1)
* Has cardiovascular disease, diabetes mellitus, Cushing's Disease, hematological malignancy, chronic mucocutaneous candidiasis or atopy
* Is pregnant or is a nursing mother
* Is a woman of child bearing potential who is not using an adequate form of contraception (or abstinence)
* Is < 19 years of age
* Suffers from a condition, which, in the opinion of the medical investigator, would compromise his/her safety

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Evidence of fungicidal activity as confirmed by mycological culture or microscopic evaluation and improvement in Clinical Symptom Severity Score | Day 12 or Day 26

SECONDARY OUTCOMES:
Incidence of adverse events | Duration of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada